CLINICAL TRIAL: NCT03884374
Title: Pain Relief for OsteoArthritis Through Combined Treatment (PROACT)
Acronym: PROACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201900232 -N; R37AG033906 (NIH); OCR20408 (Other: UF OnCore)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Adults (half AA, half NHW) with knee OA will be randomized to one of four conditions created by crossing Real tDCS vs. Sham tDCS with Focused BAT vs. Standard BAT
Who Masked: Participant, Investigator
Masking Description: Participants will be block randomized with stratification for site, sex, and race in double blind fashion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham/Sham (Experimental): Standard Breathing and Attention Training (BAT): Standard BAT intervention will incorporate most of the general aspects of the Focused BAT intervention but without the specific instructions related to mindfully attending to the breath in a non-evaluative manner.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham stimulation procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA (30s ramp up/down) of stimulation at the beginning of the session.
  Interventions: Behavioral: Standard Breathing and Attention Training (BAT); Device: Sham Transcranial Direct Current Stimulation (tDCS)
- Sham/Active (Experimental): Standard Breathing and Attention Training (BAT): Standard BAT intervention will incorporate most of the general aspects of the Focused BAT intervention but without the specific instructions related to mindfully attending to the breath in a non-evaluative manner.
  Transcranial Direct Current Stimulation (tDCS): A Soterix 1x1 Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two bicarbon rubber electrodes encased in saline-soaked sponges
  Interventions: Behavioral: Standard Breathing and Attention Training (BAT); Device: Transcranial Direct Current Stimulation (tDCS)
- Active/Sham (Experimental): Focused Breathing and Attention Training (BAT): Participants will receive mindfulness-based mental training regimen to independently practice mindfulness meditation.
  Sham Transcranial Direct Current Stimulation (tDCS): Sham stimulation procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA (30s ramp up/down) of stimulation at the beginning of the session.
  Interventions: Behavioral: Focused Breathing and Attention Training (BAT); Device: Sham Transcranial Direct Current Stimulation (tDCS)
- Active/Active (Experimental): Focused Breathing and Attention Training (BAT): Participants will receive mindfulness-based mental training regimen to independently practice mindfulness meditation.
  Transcranial Direct Current Stimulation (tDCS): A Soterix 1x1 Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two bicarbon rubber electrodes encased in saline-soaked sponges
  Interventions: Behavioral: Focused Breathing and Attention Training (BAT); Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Behavioral: Focused Breathing and Attention Training (BAT) — Participants will receive mindfulness-based mental training regimen to independently practice mindfulness meditation.
  Arms: Active/Active; Active/Sham
Behavioral: Standard Breathing and Attention Training (BAT) — Standard BAT intervention will incorporate most of the general aspects of the Focused BAT intervention but without the specific instructions related to mindfully attending to the breath in a non-evaluative manner.
  Arms: Sham/Active; Sham/Sham
Device: Transcranial Direct Current Stimulation (tDCS) — A Soterix 1x1 Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two bicarbon rubber electrodes encased in saline-soaked sponges
  Other Names: Soterix 1x1 Clinical Trials Direct Current Stimulator
  Arms: Active/Active; Sham/Active
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham stimulation procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA (30s ramp up/down) of stimulation at the beginning of the session.
  Arms: Active/Sham; Sham/Sham

SUMMARY:
This mechanistic clinical trial proposes to test whether a five-day course of mindfulness meditation training (MMT) and tDCS, and their combination, can enhance pain modulatory balance and pain-related brain function, reduce clinical pain, among African Americans and non-Hispanic whites with knee osteoarthritis (OA). This approach will provide evidence that targeting stress and pain-related brain function will reduce OA-related pain and ethnic group differences therein.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral symptomatic knee OA based on American College of Rheumatology Clinical criteria
* Participant reports primary ethnic/race group as either African American or non-Hispanic white

Exclusion Criteria:

* Actively symptomatic systemic rheumatic disease/condition (e.g. rheumatoid arthritis, systemic lupus erythematosus), or fibromyalgia that results in pain outside the knee that is equal to or worse than the participant's knee pain.
* A history of clinically significant surgery to the index knee.
* Daily use of opioids. We will exclude patients using opioids daily as both continued use and temporary withdrawal from these medications this could affect pain perception and response to interventions. Other medications being used will be recorded and controlled in statistical analyses as needed.
* Use of some centrally acting sodium channel blockers, calcium channel blockers and NMDA receptor antagonists, because some of these medications can block tDCS effects. Other medications can potentially influence response to tDCS (e.g. SSRIs, beta-blockers); therefore, consistent with recent recommendations (2), we will assess use of these medications and include them as covariates in our statistical models.
* Uncontrolled hypertension (i.e. SBP/DBP of > 150/95) or unstable or activity limiting cardiovascular or peripheral arterial disease. These exclusions are in place primarily for safety reasons, because the cold pressor task represents a cardiovascular challenge. However, uncontrolled hypertension can also affect pain perception, which is another reason for excluding these individuals.
* Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy) or evidence of previous brain injury, including stroke and traumatic brain injury.
* Serious psychiatric disorder requiring hospitalization within the past 12 months or characterized by active suicidal ideation.
* Current substance use disorder or history of hospitalization for treatment of substance use disorder.
* Diminished cognitive function that would interfere with understanding of study procedures.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Fillingim, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 317 signed consent and 251 were randomized to one of the 4 study arms. 66 people were found to be ineligible or chose not to be in the study. This is a result of additional screening being conducted after consent was obtained.
Period: Overall Study
Arm/Group | Sham/Sham | Sham/Active | Active/Sham | Active/Active
Started | 63 | 61 | 64 | 63
Completed | 63 | 61 | 64 | 63
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham/Sham | Sham/Active | Active/Sham | Active/Active | Total
Number analyzed (Participants) | 63 | 61 | 64 | 63 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 36 | 43 | 169
  >=65 years | 18 | 16 | 28 | 20 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (9.2) | 60.6 (8.9) | 63.4 (8.2) | 60.1 (9.3) | 61.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 43 | 43 | 168
  Male | 20 | 22 | 21 | 20 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 63 | 61 | 64 | 63 | 251
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 30 | 31 | 32 | 33 | 126
  White | 33 | 30 | 32 | 30 | 125
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 63 | 63 | 251

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
Description: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): 26 question index to assess knee OA pain (0-20 scale), function (0-68 scale), and stiffness (0-8 scale). The total WOAMC score is the sum of the 3 sub scales for a total score range from 0-96. Change in total WOMAC score = V7 total WOMAC score - Baseline (pre-intervention) total WOMAC score. The lower change scores represents improvement in pain, movement, and stiffness.
Time Frame: Visit 1-Baseline prior to intervention and Visit 7 which is about 1 month after baseline visit and study intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham/Sham | Sham/Active | Active/Sham | Active/Active
Number analyzed (Participants) | 63 | 61 | 64 | 63
units on a scale | -6.5 (11.3) | -3.8 (13.5) | -7.4 (12.1) | -6.3 (15)

ADVERSE EVENTS:
Time Frame: about 3 months
Arm/Group | Sham/Sham | Sham/Active | Active/Sham | Active/Active
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/61 | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/61 | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 2/63 | 3/61 | 4/64 | 2/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham/Sham (N=63) | Sham/Active (N=61) | Active/Sham (N=64) | Active/Active (N=63)
Blurry vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pain (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03884374/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03884374/ICF_000.pdf